CLINICAL TRIAL: NCT06339645
Title: The Correlation of Safety and Effectiveness Between Intravesical Platelet-rich Plasma Injection in Patients With Interstitial Cystitis/Bladder-A Retrospective Study
Brief Title: Intravesical Platelet-rich Plasma Injection in Patients With Interstitial Cystitis/Bladder-A Retrospective Study
Status: Not yet recruiting | Type: Observational
Sponsor: Hualien Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Wan Ru Yu, PI, Hualien Tzu Chi General Hospital
Other Study IDs: P00003121
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Safety and Effectiveness Between Intravesical Platelet-rich Plasma Injection in Patients With Interstitial Cystitis/Bladder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PRP — Patients who meet all eligibility requirements for entry into the study of intravesical PRP injection

SUMMARY:
The correlation of safety and effectiveness between intravesical platelet-rich plasma injection in patients with interstitial cystitis/bladder-A retrospective study to evaluate the correlation of safety and effectiveness between intravesical platelet-rich plasma injection of IC/BPS, with age of at least 20-84 years old in Taiwan of either sex with IC/BPS symptoms and proven of IC by cystoscopic hydrodistention. Patients who meet all eligibility requirements for entry into the study of intravesical PRP injection.

DETAILED DESCRIPTION:
Introduction: Interstitial cystitis/bladder pain syndrome (IC/BPS) is a chronic inflammatory disease of the bladder characterized by symptoms such as frequency, urgency, nocturia, and lower abdominal pain. Despite being recognized for a hundred years, there has not been a definitive treatment method that can completely eliminate bladder inflammation. Various methods have been attempted, including bladder hydrodistention, anti-inflammatory drugs, steroid injections, and the use of bladder epithelial protectants such as Hyaluronic Acid. In recent years, the use of intravesical injection of botulinum toxin for the treatment of IC/BPS has emerged; however, none of these methods have achieved the goal of long-term cure. Therefore, achieving remission of interstitial cystitis has been a persistent goal for urologists.

Platelet-rich plasma (PRP) therapy has emerged as a novel treatment modality in the past one to two decades, widely used for degenerative joint diseases and muscle injuries. This therapy involves extracting high concentrations of platelets mixed with serum from the patient's own blood, excluding red and white blood cells, and injecting this high-concentration platelet serum into the affected area. This exploits the various growth factors and cytokines abundant in platelets to promote wound healing and reduce chronic inflammation. PRP has shown promising results in many sports injuries and degenerative joint diseases over the past decade. As PRP is derived from the patient's own blood, it does not induce allergic reactions or produce any side effects.

PRP has been previously shown to effectively improve epithelial dysfunction and chronic inflammation in IC/BPS. We hope PRP injection can gradually eliminate inflammation within the bladder, and its various growth factors can facilitate the repair of damaged bladder epithelium. If this treatment proves effective, it could offer a better therapeutic option for many patients suffering from bladder symptoms due to interstitial cystitis.

Several patients have been enrolled since the initiation of clinical trials using intravesical injection of platelet-rich plasma for bladder treatment in 2016. However, data collection has been limited to single clinical trial studies. PRP has gradually become a routine treatment for patients with IC/BPS. Therefore, this study aims to comprehensively review the medical records of all patients who have received bladder PRP injections to clarify and understand the basic information and clinical examination data of patients with interstitial cystitis who have received bladder PRP injections from the past to the present.

Aim: This study also aims to understand interstitial cystitis further and investigate the safety and efficacy of bladder PRP injections for patients with interstitial cystitis.

Materials and Methods:

This retrospective study enrolled the patients who received intravesical PRP injection treatments in patients with IC/BPS from 2016/1/1 to 2023/10/21. We used the chart review and questionnaire collection, analyzed the patients' characteristics including age, gender, IC symptoms, and pain severity, and also collected anxiety severity all in the chart. Also, the voiding diary, maximum bladder capacity, urine biomarkers, and glomerulation grade were analyzed.

Assessment: The patients will be investigated using the chart review for the voiding diary (for frequency nocturia episodes per day), ICSI, IC problem index (ICPI), Numerical Rating Scale (NRS) of pain, patient perception of bladder condition (PPBC), global response assessment (GRA), maximal flow rate (Qmax), voided volume (Vol), and post-void residual urine (PVR) volume measurement at baseline and after treatment. Urine samples will also be obtained for urinary biomarkers determination at baseline and after different therapy.

ELIGIBILITY:
Inclusion Criteria:

* NIDDK criteria diagnostic IC/BPS, and received the intravesical PRP injection before

Exclusion Criteria:

1. non-IC/BPS patients
2. psychological disease was diagnosed
3. non-NIDDK criteria (Hunner's ulcer type)
4. Under-primary or illiterate respondents
5. patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow up
6. Patients with bladder outlet obstruction on enrollment
7. Patients with post-void residual > 150ml
8. Patients with an uncontrolled confirmed diagnosis of acute urinary tract infection
9. Patients have laboratory abnormalities at screening
10. Patients who cannot used urinary catheter to treat.
11. Female patients who are pregnant, lactating, or childbearing potential without contraception.
12. Patients with any other serious disease considered by the investigator not in the condition to enter the trial
13. Patients cannot record the voiding diary

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with age of at least 20-84 years old in Taiwan of either sex with IC/BPS symptoms and proven of IC by cystoscopic hydrodistention
Sampling Method: Non-Probability Sample
Enrollment: 658 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-05-22 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Global response assessment (GRA) | 6 months
  satisfaction by the patient (categorized into -3, -2,-1, 0, +1, +2, +3, indicating markedly worse to markedly improved ) after the treatment day

CONTACTS AND LOCATIONS:
Overall Officials: Wan Ru Yu, Principal Investigator — Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien, Taiwan,
Locations (1):
- Wan Ru Yu, Hualien City, Outside U.S./Taiwan, Taiwan

REFERENCES:
- [Derived] Yu WR, Kuo HC. Functional bladder capacity can reflect the bladder condition and treatment outcome in patients with interstitial cystitis/bladder pain syndrome. World J Urol. 2026 Jan 17;44(1):101. doi: 10.1007/s00345-025-05937-2. No abstract available. PMID 41546691